CLINICAL TRIAL: NCT06086236
Title: Effects of Transcutaneous Auricular Vagus Nerve Stimulation on Basic Autonomic Nervous System Activity
Brief Title: Vagus Nerve Stimulation Effects on Autonomic Nervous System Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Alper Percin, Principal Investigator, Bahçeşehir University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AP00013
Record Dates: First submitted 2023-10-06; First posted 2023-10-17 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Vagus Nerve Stimulation
Keywords: Vagus Nerve Stimulations; Diastolic Pressure; Pulse Rate; Systolic Pressure

STUDY DESIGN:
Intervention Model Description: After the participants were included in the study, heart rate variability was measured and divided into 4 groups according to PNS and SNS indexes.
Who Masked: Outcomes Assessor
Masking Description: The evaluations were carried out by the second researcher
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PNS Index<-2 and SNS Index>2 (Experimental): Participants with Parasympathetic Nervous System (PNS) and Sympathetic Nervous System (SNS) Indexes values ''PNS<-2, SNS>2'' according to the results of heart rate variability measurements were included in this group. Then bilateral transcutaneous auricular vagus nerve stimulation was performed.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- PNS Index<-2 and SNS Index<2 (Experimental): Participants with Parasympathetic Nervous System (PNS) and Sympathetic Nervous System (SNS) Indexes values ''PNS<-2, SNS<2'' according to the results of heart rate variability measurements were included in this group. Then bilateral transcutaneous auricular vagus nerve stimulation was performed.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- PNS Index>-2 and SNS Index>2 (Experimental): Participants with Parasympathetic Nervous System (PNS) and Sympathetic Nervous System (SNS) Indexes values ''PNS>-2, SNS>2'' according to the results of heart rate variability measurements were included in this group. Then bilateral transcutaneous auricular vagus nerve stimulation was performed.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation
- PNS Index>-2 and SNS Index<2 (Experimental): Participants with Parasympathetic Nervous System (PNS) and Sympathetic Nervous System (SNS) Indexes values ''PNS>-2, SNS<2'' according to the results of heart rate variability measurements were included in this group. Then bilateral transcutaneous auricular vagus nerve stimulation was performed.
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Through a special Ear set, bilateral Transcutaneous Auricular Vagus Nerve Stimulation was applied to all participants for 20 minutes.

SUMMARY:
Transcutaneous Auricular Vagus nerve stimulation may be successful in cardiac modulation because of the cardiac connections of the vagal nerve. Therefore, in order to observe the cardiac effects, it was analysed the changes in pulse rate, systolic and diastolic blood pressure after transcutaneous auricular vagus nerve stimulation application.

DETAILED DESCRIPTION:
Participants were divided into four groups (Figure 1) according to PNS and SNS indexes as Group 1 (PNS index <-2, SNS index >+2), Group 2 (PNS index <-2, SNS index <+2), Group 3 (PNS index >-2, SNS index >+2), Group 4 (PNS index >-2, SNS index <+2). Participants were assessed with blood pressure, pulse rate and HRV before and after taVNS stimulation. Sympathetic nervous system (SNS) index and parasympathetic nervous system (PNS) index values were assumed to be between -2 and +2 (95%) in the normal population according to Kubios software, and the grouping method was based on this situation.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years old.
* No previous vagus nerve stimulation

Exclusion Criteria:

* Using of any drug, alcohol or smoking.
* Pregnancy.
* Known history of acute or chronic illness.
* Being in the post or peri-menopausal stage.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-10 (Actual)

PRIMARY OUTCOMES:
Pulse Rate | Up to 6 Months
  The pulse rate of the participants was measured with an electronic blood pressure monitor.
Systolic Blood Pressure | Up to 6 Months
  The systolic blood pressure of the participants was measured with an electronic blood pressure monitor.
Diastolic Blood Pressure | Up to 6 Months
  The diastolic blood pressure of the participants was measured with an electronic blood pressure monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Alper Perçin, Ph.D., Principal Investigator — Igdir University
Locations (1):
- Igdir University, Iğdır, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It is not preferred to share the data until the study is published.

REFERENCES:
- [Background] Wang Y, Li SY, Wang D, Wu MZ, He JK, Zhang JL, Zhao B, Hou LW, Wang JY, Wang L, Wang YF, Zhang Y, Zhang ZX, Rong PJ. Transcutaneous Auricular Vagus Nerve Stimulation: From Concept to Application. Neurosci Bull. 2021 Jun;37(6):853-862. doi: 10.1007/s12264-020-00619-y. Epub 2020 Dec 23. PMID 33355897
- [Background] Ben-Menachem E, Revesz D, Simon BJ, Silberstein S. Surgically implanted and non-invasive vagus nerve stimulation: a review of efficacy, safety and tolerability. Eur J Neurol. 2015 Sep;22(9):1260-8. doi: 10.1111/ene.12629. Epub 2015 Jan 23. PMID 25614179
- [Background] Milby AH, Halpern CH, Baltuch GH. Vagus nerve stimulation for epilepsy and depression. Neurotherapeutics. 2008 Jan;5(1):75-85. doi: 10.1016/j.nurt.2007.10.071. PMID 18164486
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Borovikova LV, Ivanova S, Zhang M, Yang H, Botchkina GI, Watkins LR, Wang H, Abumrad N, Eaton JW, Tracey KJ. Vagus nerve stimulation attenuates the systemic inflammatory response to endotoxin. Nature. 2000 May 25;405(6785):458-62. doi: 10.1038/35013070. PMID 10839541
- [Background] Sinniger V, Pellissier S, Fauvelle F, Trocme C, Hoffmann D, Vercueil L, Cracowski JL, David O, Bonaz B. A 12-month pilot study outcomes of vagus nerve stimulation in Crohn's disease. Neurogastroenterol Motil. 2020 Oct;32(10):e13911. doi: 10.1111/nmo.13911. Epub 2020 Jun 8. PMID 32515156
- [Background] Sigurdsson HP, Raw R, Hunter H, Baker MR, Taylor JP, Rochester L, Yarnall AJ. Noninvasive vagus nerve stimulation in Parkinson's disease: current status and future prospects. Expert Rev Med Devices. 2021 Oct;18(10):971-984. doi: 10.1080/17434440.2021.1969913. Epub 2021 Sep 8. PMID 34461787
- [Background] Badran BW, Dowdle LT, Mithoefer OJ, LaBate NT, Coatsworth J, Brown JC, DeVries WH, Austelle CW, McTeague LM, George MS. Neurophysiologic effects of transcutaneous auricular vagus nerve stimulation (taVNS) via electrical stimulation of the tragus: A concurrent taVNS/fMRI study and review. Brain Stimul. 2018 May-Jun;11(3):492-500. doi: 10.1016/j.brs.2017.12.009. Epub 2017 Dec 29. PMID 29361441
- [Background] Redgrave J, Day D, Leung H, Laud PJ, Ali A, Lindert R, Majid A. Safety and tolerability of Transcutaneous Vagus Nerve stimulation in humans; a systematic review. Brain Stimul. 2018 Nov-Dec;11(6):1225-1238. doi: 10.1016/j.brs.2018.08.010. Epub 2018 Aug 23. PMID 30217648
- [Background] Sclocco R, Garcia RG, Kettner NW, Isenburg K, Fisher HP, Hubbard CS, Ay I, Polimeni JR, Goldstein J, Makris N, Toschi N, Barbieri R, Napadow V. The influence of respiration on brainstem and cardiovagal response to auricular vagus nerve stimulation: A multimodal ultrahigh-field (7T) fMRI study. Brain Stimul. 2019 Jul-Aug;12(4):911-921. doi: 10.1016/j.brs.2019.02.003. Epub 2019 Feb 10. PMID 30803865